CLINICAL TRIAL: NCT02843620
Title: Randomized Double-blind, Placebo Controlled Study to Asses the Efficacy and Safety of a Native Collagen Food Supplement on Joint Function, Ultrasound Evolution and Quality of Life of Adults With Moderate Knee Pain
Brief Title: Efficacy and Safety of b-2Cool on Adults With Joint Discomfort
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment not started
Sponsor: Bioiberica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRJ290
Record Dates: First submitted 2016-07-19; First posted 2016-07-26 (Estimated); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Joint Discomfort
Keywords: Native Collagen; Joint; Joint Discomfort

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): The placebo arm will take a pill each day containing only excipients
  Interventions: Other: Placebo
- b-2Cool (Experimental): The b-2Cool arm will take a pill each day containing 40 mg of b-2Cool and excipients
  Interventions: Dietary Supplement: b-2Cool

INTERVENTIONS:
Dietary Supplement: b-2Cool — b-2Cool® is native type II collagen extracted from chicken sternums
  Arms: b-2Cool
Other: Placebo — Excipients only
  Arms: Placebo

SUMMARY:
This study evaluates the effects of 40 mg of b-2Cool, a food supplement rich in native type-II collagen, on healthy adults with joint discomfort. Half of the participants will receive the b-2Cool containing supplement while the other half will receive a placebo pill.

DETAILED DESCRIPTION:
Previous studies had shown the efficacy of the intake of native collagen to relieve pain in healthy patients with joint discomfort.

Native collagen is detected in the gut's Peyer's patches and, thanks to a mechanism known as oral tolerisation, reduces the autoimmune attack to joints' collagen improving joint function and pain.

Oral tolerance consists of two phases of immune response: the maintenance of homeostasis and the suppression of immune responses mediated by Ag-specific regulatory T cells. T-cells detect the epitopes of type-II collagen in the gut and suppress the immune response against bodily type-II collagen. Then, these regulatory T cells generated in the gut are presumed to migrate to a local microenvironment where a protein analogous to the orally dosed antigen resides, in this case type-II collagen. Upon reactivation in a new microenvironment, regulatory cells will suppress ongoing inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 40 and 75 years old.
* Subject who suffers mild joint discomfort (value between 3 and 5 VAS scale for a minimum of 6 months).
* Subject that after reading and understanding the study's protocol has provided written informed consent to participate in the study.
* Subjects willing to keep stable eating and activity patterns during the duration of the study.
* Subjects who use other therapies for joint discomfort, such as exercise, heat / cold, joint protection and physiotherapy / occupational therapy agree to follow the treatments avoiding changes in the frequency or intensity of them and reporting them at baseline and during follow-ups.
* Subjects agree not start any new therapy during the study period.
* Subjects who have lateral or longitudinal knee synovial effusion according to the index OMERACT (Outcome Measures in Rheumatology) .

Exclusion Criteria:

* Active rheumatoid arthritis, diagnosed osteoarthritis or any other inflammatory arthritic condition that researchers consider non appropriate.
* Being pregnant or lactating.
* Be waiting for joint surgery or major surgery in the next 8 months
* Joint injury in the last 4 months in the area osteoarthritis-affected (i.e. meniscal tear)
* Having underwent reconstructive surgery on the cartilage of the affected knee
* Background of peptidic ulcer and other symptomatic/active disorders of the intestinal tract that may interfere with product under evaluation .
* History of congestive heart failure,
* Allergy to chicken or other ingredients in the product
* Anticipated problems with product consumption
* High alcohol consumption (> 2 drinks per day)
* History of psychiatric disorders that may impede the ability of subjects to give written informed consent
* Failure to comply with washout periods before the start of the study.
* Paracetamol intake 24 hours before randomization
* The subject does not want to stop taking medication in addition to the study medication (for arthritis or other pain) or not to take other types of medication for the treatment of osteoarthritis pain
* Other conditions that, in the opinion of the principal investigator adversely affect the subject's ability to complete the study or its measures

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07 (Estimated); Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of ultrasonographic assessment of synovial effusion | 0, 6, 12 and 24 weeks

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) pain evaluation | 0, 6, 12 and 24 weeks
WOMAC Functional assesment | 0, 6, 12 and 24 weeks
Subjective evaluation of quality of life | 0, 6, 12 and 24 weeks
  Patients will report some aspects of their Quality of life through Visual analogic scales
Collagen degradation markers in urine | 0, 12 and 24 weeks
Patient's satisfaction | 6, 12 and 24 weeks
  Patient satisfaction will be evaluated using a subjective questionnaire
Rescue medication consumption | Every 2 weeks for 24 weeks
Adverse events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Möller, Dr., Principal Investigator — Instituto Poal de Reumatología

IPD SHARING:
Plan to Share IPD: Undecided